CLINICAL TRIAL: NCT01454492
Title: The Relationship Between Allergic Rhinitis and Geographic Tongue
Acronym: AR-GT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH-3485
Record Dates: First submitted 2011-10-04; First posted 2011-10-19 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Allergic Rhinitis; Geographic Tongue
Keywords: Allergy rhinitis; Geographic tongue
MeSH Terms: conditions — Rhinitis, Allergic; Glossitis, Benign Migratory

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Allergy rhinitis: Allergy rhinitis patients group
- Non- Allergy rhinitis: Non- Allergy rhinitis patients group

SUMMARY:
Allergic rhinitis is a complex chronic inflammatory disease, it always presents with nasal obstruction, nasal itching, sneezing and runny nose. Whether in adults or children, rhinitis is a complex disease. The prevalence of allergic rhinitis in Taiwan is about 24-29%. Taiwan is a developing country. It is a hot and humid country. In developing countries, industrialization, air pollution makes the constantly increasing number of patients with rhinitis. Penghu in 1994 for children aged 7 to 14 by the study found that among 7599 people, 1766 people have allergic rhinitis, about 23.2%. Allergic rhinitis is a complex chronic disease. So, it become a diagnostic challenge, its prevalence always underestimated. The prevalence of rhinitis has increased in recent years. The phenomenon of underestimate is caused by variety of personal and environmental factors. Allergic rhinitis had increased direct and indirect social and economic burden.

Geographic tongue is a benign tongue performance. Geographic tongue has been reported their relevance to allergy. Geographic tongue is a chronic tongue situation. The causes of geographic tongue still remains unknown. Allergic rhinitis is a diagnostic challenge to clinicians. The investigators hope that geographic tongue could play a role in the diagnostic of allergic rhinitis. The prevalence of geographic tongue in the United States is about 1.8%, white Americans and Mexicans have a higher incidence rate. This study will investigate the relevance between allergic rhinitis and geographic tongue. The investigators will analyze the relevant gender, age, severity of inspection reports. The research results wound provide an important reference to the diagnosis of allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* rhinitis and non-rhinitis patients
* willing to complete the study
* no limitation of tongue movement

Exclusion Criteria:

* more than 90 years old or younger than 20 years old
* unable to complete the study

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: Allergy rhinitis Group 2: Non-allergy rhinitis
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-03 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | 8th month

CONTACTS AND LOCATIONS:
Overall Officials: CJ Tai, M.D., Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan, Taiwan

REFERENCES:
- [Result] Miloglu O, Goregen M, Akgul HM, Acemoglu H. The prevalence and risk factors associated with benign migratory glossitis lesions in 7619 Turkish dental outpatients. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009 Feb;107(2):e29-33. doi: 10.1016/j.tripleo.2008.10.015. PMID 19138635
- [Result] Reamy BV, Derby R, Bunt CW. Common tongue conditions in primary care. Am Fam Physician. 2010 Mar 1;81(5):627-34. PMID 20187599
- [Result] Masferrer E, Jucgla A. Images in clinical medicine. Geographic tongue. N Engl J Med. 2009 Nov 12;361(20):e44. doi: 10.1056/NEJMicm0810145. No abstract available. PMID 19907039
- [Result] Shulman JD, Carpenter WM. Prevalence and risk factors associated with geographic tongue among US adults. Oral Dis. 2006 Jul;12(4):381-6. doi: 10.1111/j.1601-0825.2005.01208.x. PMID 16792723
- [Result] Ugar-Cankal D, Denizci S, Hocaoglu T. Prevalence of tongue lesions among Turkish schoolchildren. Saudi Med J. 2005 Dec;26(12):1962-7. PMID 16380783